CLINICAL TRIAL: NCT02376439
Title: Non-shared Environments and Discordance of Obesity in Adolescent Sibilngs
Brief Title: Discordance of Obesity in Adolescent Sibilngs
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 1087494-1-54072
Record Dates: First submitted 2014-07-18; First posted 2015-03-03 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: siblings; overweight; adolescent
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Siblings: Siblings will consume four test meals after 4 different exposures, including two types of koolaid, a control and a smell condition.
  Interventions: Other: Kool-aid

INTERVENTIONS:
Other: Kool-aid — Participant drank two different types of kool-aid (sugar free and regular)

SUMMARY:
This research studies the energy balance behaviors (usual eating, physical activity, sedentary) and non-shared experiences of siblings discordant for weight (one sibling is lean the other is overweight).

DETAILED DESCRIPTION:
This research studies the energy balance behaviors (usual eating, physical activity, sedentary) and non-shared experiences of siblings discordant for weight (one sibling is lean the other is overweight). To accomplish this, siblings attend four laboratory sessions where they consume one of two types of kool-aid, smell the pizza, or rest quietly. Siblings then eat a dinner meal. Siblings also wear an activity monitor for one week and record their physical activity and sedentary activities in a habit book.

ELIGIBILITY:
Inclusion Criteria:

* between 13-17 years old
* Have discordant same gender sibling (one is below 70th percentile, one is above 85th percentile
* Speak/read English
* Moderate or greater liking of study foods

Exclusion Criteria:

* No current diagnosis of a psychiatric or eating disorder.
* No dieting, dietary restrictions, or allergies that would interfere with study participation.
* No medications or conditions that could influence taste or appetite.
* No health concern or physical disability that would limit participation in physical activity.
* No endocrine or central nervous system disorder that could produce overweight.
* No current use of tobacco or nicotine products by the adolescent siblings.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Forty-eight sibling pairs (24 pairs of boys and 24 pairs of girls, 96 total adolescents) age 13 to 17 years who are discordant for overweight/obesity will be studied to assess potentially modifiable non-shared experiences within and outside the family environment that alter energy balance behaviors and contribute to adolescent overweight. We will also measure the height and weight of up to 3 of their best friends.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Internal and external satiety calories consumed | Calories consumed are measured at week 1, week 2, week 3 and week 4.
  Calories consumed during ad libitum meals are measured after consumption of a high energy dense preload and a low energy dense preload and also after an external cue (smell) and a control condition.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Epstein, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States